CLINICAL TRIAL: NCT00817739
Title: Intermittent Hormonal Therapy With Leuprorelin (3.75 mg SR) and Flutamide in the Treatment of Stage D2 or Tx Nx M1 ≠ M1a Metastatic Cancer of the Prostate
Brief Title: Intermittent Hormonal Therapy With Leuprorelin and Flutamide in the Treatment of Stage D2 or TxNxM1b,c
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAP IIb/95/022 - EC210; U1111-1169-6769 (Registry Identifier: WHO)
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Prostatic Neoplasms
Keywords: Drug therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Flutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Therapy (Active Comparator): Continuous complete androgen suppression therapy with leuprorelin 3.75 mg sustained release (SR), injection, subcutaneously once every 28 days and flutamide, 250 mg, tablet, orally thrice daily until there are signs of disease progression.
  Interventions: Drug: Leuprorelin; Drug: Flutamide
- Intermittent therapy (Experimental): Intermittent complete androgen suppression therapy starting at randomization with interruption of treatment given in the induction period until PSA levels reach >=10 ng/mL or other signs of progression appear. Upon treatment resumption, leuproreline 3.75 mg SR, injection, subcutaneously once every 28 days and flutamide 250 mg, tablet, orally thrice daily, until PSA levels are <normal (that is, <4 ng/mL) and no signs of disease progression appear. The intermittent therapy will be continued similarly until the study end or the appearance of signs of disease progression under treatment.
  Interventions: Drug: Leuprorelin; Drug: Flutamide

INTERVENTIONS:
Drug: Leuprorelin — Leuprorelin injection
Drug: Flutamide — Flutamide tablets

SUMMARY:
This study is aimed at evaluating the effects of intermittent hormonal treatment with complete androgen suppression (Leuprorelin 3.75 milligram [mg] sustained release [SR] and Flutamide) in patients presenting with stage D2 or Tx Nx M1 ≠ M1a metastatic prostrate cancer, with a prostate specific antigen (PSA) level 5-fold higher than normal (PSA greater than or equal to [≥] 20 nanogram per milliliter [ng/mL], as quantitated by the Hybritech radioimmunoassay) and with a subsequent decline to normal (PSA less than [<] 4 ng/mL) during the initial 6 months of induction treatment. The results will be compared with those obtained after continuous hormonal therapy with complete androgen suppression.

DETAILED DESCRIPTION:
This is an open, comparative, randomized (1:1), multicenter, European (France, Germany, Czech Republic, Slovakia and Bulgaria), Phase 2B study on parallel groups of patients presenting with metastatic prostate cancer (stage D2 or Tx Nx M1 ≠ M1a), with a PSA level ≥ 5-fold higher than normal (that is PSA ≥ 20 ng/mL, as quantitated by the Hybritech radioimmunoassay) which return to normal within 6 months after the initiation of total androgen blockade therapy with leuprorelin 3.75 mg SR and flutamide. It will involve 314 preselected patients.

A minimum of 180 eligible patients are required for this study. Selected patients will be randomized centrally in two parallel groups at study entry. This phase 2B study will enable evaluation of a high number of patients by direct comparison with conventional administration. The study comprises of two therapeutic phases:

* A 6 month induction phase with complete androgen suppression by leuprorelin 3.75 mg SR and flutamide. This phase involves patients meeting the preselection criteria.
* A data processing run per complete androgen suppression according to two methods, continuous or intermittent, for the patients satisfying the criteria of selection of the study and which will thus be randomized.

The selected patients will be randomized in two parallel groups at the time of inclusion:

* Group A patients will receive a continuous complete androgen suppression therapy by leuprorelin 3.75mg SR and flutamide, until the appearance of signs of disease progression or study end.
* Group B patients will receive an intermittent complete androgen suppression therapy by leuprorelin 3.75 mg SR and flutamide, until the study end or the appearance of signs of disease progression under treatment.

Group A patients will be routinely followed-up on a 3-month basis until there are signs of disease progression. Group B patients (intermittent therapy) will be monitored every 3 months during on-treatment periods under the same conditions as described for group A.

The 3-month clinical follow-up will be same during off-treatment periods, but if PSA increases to ≥10 ng/mL the patient must be contacted to schedule a prompt special visit in order to reinstitute hormonal therapy. Subsequent visits will be scheduled on a 3-month basis from the time of the special visit. Special visits will be the same as routine consultations, except that the laboratory tests will not be redone.

When on-therapy tumor progression will be documented, every 6 months the investigators will note all treatments administered to patients until death (while specifying the cause of death).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic cancer of the prostate (stage D2 or Tx Nx M1 ≠ M1a) with measurable bone or visceral (lung, liver, etc.) metastases (radiographic conformation was necessary in the event of a questionable bone scan detection in conjunction with only slightly elevated PSA levels [at least 20 ng/mL or less than or equal to 50 ng/mL]). The prostatic carcinoma could have been diagnosed at an earlier stage and treated without castration.
* Metastatic cancer of the prostate requiring first-line therapy.
* Pre-assessment PSA 5-fold or higher than the standard level set by the central laboratory, that is, PSA greater than or equal to (≥) 20 ng/mL as quantitated by the Hybritech radioimmunoassay (normal is less than [<] 4 ng/mL).
* ECOG performance status of no more than 2.
* Normal testosterone levels according to the central laboratory standards.
* Aspartate transaminase (AST) and alanine transaminase (ALT) < 2.25-fold higher than the standard levels set by the central laboratory (except when liver metastases were present).
* Anticipated life expectancy greater than 9 months.
* Written informed consent given to participate and collaborate in the study. Inclusion Criteria for Continuous or Intermittent Treatment Phase
* Subjects who meet the pre-assessment criteria and who has PSA < 4 ng/mL after 6 months of induction therapy.

Exclusion Criteria:

* Subject refuse to sign the informed consent form or is likely to be uncooperative or not to comply with the obligations set out in the study protocol.
* Subject has received prior hormonal (and neoadjuvant) treatment prompting medical castration (estrogens, hormone-releasing hormone agonists, androgens) or has undergone surgical castration.
* Subject has undergone bilateral suprarenalectomy or hypophysectomy.
* Subject had another cancer (except basiloma) with the past 5 years.
* Subject has serious unstable progressive disease (renal, hepatic, cardiovascular, psychological, etc).
* Subject is receiving or has received another experimental treatment within 3 months prior to inclusion.

Exclusion Criteria for Continuous or Intermittent Treatment Phase

-Subjects who met the pre-assessment criteria and who, after 6 months of induction therapy, had PSA ≥ 4 ng/mL and/or on-treatment signs of disease progression.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 1996-12; Primary Completion 2005-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Median Overall Survival | Randomization (Month 6) up to Week 396 after randomization
  Median Overall survival is defined as the number of days from date of inclusion to the date of death. For subjects who do not die, survival will be censored at the date of last contact.
Median Progression-Free Survival | Randomization (Month 6) up to Week 396 after randomization
  Median Progression Free Survival=time from date of inclusion to date of first documentation of progressive disease (death, biological progression, clinical progression). Biological progression: date of the first PSA increase after the nadir and greater than or equal to (≥) 4 ng/mL under treatment. Clinical progression: date of appearance of the clinical sign of progression under treatment. Clinical signs of progression are: 1. Appearance of marked increase of bone pain or appearance of symptoms related to disease progression (example: liver, lungs, kidneys); 2. Alteration of general health conditions related to disease progression (decrease of at least 2 degrees in the European Organization for Research and Treatment of Cancer (ECOG) performance status, weight loss of more than 10% since the last visit); 3. Anemia - drop in hemoglobin level of more than 2 gram per deciliter (g/dL) since the last visit (only if disease related).

SECONDARY OUTCOMES:
European Organization for research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) - C30 | Randomization (Month 6) up to Week 396 after randomization
  EORTC QLQ-C30: includes functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). Most questions uses 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions uses 7-point scale (1 'very poor' to 7 'Excellent'). Scores are averaged and transformed to 0-100 scale; for the 5 functional scales and the global quality-of-life scale, a higher score represents a better level of functioning. For the symptom-oriented scales and items, a higher score corresponds to a higher level of symptoms.
Change from Baseline in Subjective Clinical Efficacy (Symptomatic) | Randomization (Month 6) up to Week 396 after randomization
  Subjective clinical efficacy will be assessed using the Madsen Symptom Index and Lukacs' questionnaire. Symptoms will be assessed using visual analogue scale (VAS) in Lukacs questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MOTTET, MD, Principal Investigator — Clinique Mutualiste de Saint-Etienne